CLINICAL TRIAL: NCT06982443
Title: Mindfulness-Based Relapse Prevention and Psychophysiological Self-Regulation
Brief Title: Wellness, Alcohol, Vitals, and Emotions
Acronym: WAVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Matison McCool, Research Assistant Professor, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2407142185; K23AA031729 (NIH)
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use
Keywords: alcohol; mindfulness; harm reduction
MeSH Terms: conditions — Alcohol Drinking; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MBRP (Experimental)
  Interventions: Behavioral: Mindfulness based relapse prevention

INTERVENTIONS:
Behavioral: Mindfulness based relapse prevention — Mindfulness-based relapse prevention (MBRP) is a group-based treatment to provide individuals with skills intended to foster increased awareness of triggers, destructive habitual patterns, and "automatic" reactions to triggering experiences. Mindfulness practices in MBRP are designed to help individuals pause, observe present experience, and bring awareness to the range of choices available in every moment. Through MBRP individuals learn to respond in ways that serve them, rather than react in ways that are detrimental to their health and happiness.
  Other Names: MBRP

SUMMARY:
The goal of this clinical trial is to examine the effects of mindfulness based relapse prevention on self-regulation overtime and drinking in daily life through the use of wearable heart rate sensors during mindfulness groups and answering assessment questions 3 times per day during the course of treatment. The main questions that it aims to answer are:

1. What changes in self-regulation as measured through heart rate variability are observed during a mindfulness intervention and how do those self-regulatory changes affect drinking after treatment?
2. How do changes in heart rate variability affect drinking, craving, and negative affectivity in daily life?

Participants will:

1. Answer questions related to their mood and drinking behaviors.
2. Wear their sensors during an 8-week treatment period with 1 group per week.
3. Answer questions 3 times a day during the treatment period. 4.) Return their sensors via a pre-stamped package and answer questions about their mood and drinking behaviors 3- and 6-months after the mindfulness groups end.

DETAILED DESCRIPTION:
This study will assess the changes in self-regulation as measured through heart rate variability (HRV), that occur during the course of an 8-week mindfulness-based relapse prevention (MBRP) treatment. The investigators will use a single-group design to test the effects of MBRP on resting, reactivity, and recovery HRV. Additionally, the study will test whether changes in HRV that occur week over week during treatment can affect drinking behaviors in daily life. Individuals (n=120) who meet criteria for moderate to severe alcohol use disorder will be mailed small HRV sensors to be worn before, during, and after each MBRP group. Participants will answer questions about their functioning, alcohol use, addiction cycle domains, and mood at baseline, and at follow-up months 3 and 6.

MBRP groups will be delivered at the same time each week for 8 consecutive weeks, known as the treatment period. During the treatment period, participants will self-attach their sensors before each MBRP group, watch a brief presentation to collect resting HRV, complete their group, and watch a brief presentation after each group. During the treatment period, participants will also answer questions about their drinking, functioning, and mood 3 times a day.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Meet criteria for a moderate to severe alcohol use disorder within the previous 3-months.
3. Able to attend group meetings at the time listed on the recruitment materials.
4. Willing to wear a sensor for the 8-week intervention period and return the sensor after the immediate follow-up.
5. Have a phone/tablet/computer with internet access.
6. Be able to comprehend and consent to study requirements in English.
7. Have access to a valid U.S. mailing address for receiving the HRV sensors and reside in the United States.

Exclusion Criteria:

1. Current symptoms of psychosis or mania.
2. Have a substance use disorder requiring a higher level of care than outpatient treatment (e.g., severe alcohol use disorder requiring inpatient detoxification).
3. Have a history of pulmonary or cardiovascular disease that interferes with sensor data collection and HRV metrics (i.e., ectopic beats, arrythmia, congenital heart disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Recovery from AUD | Change from baseline to 6-month follow-up
  Recovery is a binary (yes/no) outcome defined by achieving all three of the following: (1) Remission from Diagnostic and Statistical Manual, 5th edition alcohol use disorder (AUD) based on an 11-item AUD symptom checklist (endorsing 0 or 1 item is AUD remission); (2) Cessation of heavy drinking (defined as not engaging in heavy drinking with heavy drinking defined as 4 or more drinks per occasion for females, and 5 or more drinks per occasion for males, measured by the Timeline Follow-Back); and (3) Improvements in functioning and well-being as measured by higher score on the PROMIS PROPr measure. Recovery is achieved if remission, cessation of heavy drinking, and improvements in functioning and well-being are achieved. These assessments will be delivered at Baseline, 3-month, and 6-month follow-ups.
Psychophysiological self-regulation | Change from baseline to immediate follow-up
  Psychophysiological self-regulation will be measured through three heart rate variability (HRV) domains: HRV at rest (higher RMSSD/HF-HRV indicate higher self-regulation), reactivity HRV (no change, or increases in HRV indicate less reactivity), and recovery HRV (quicker return to resting HRV indicates greater recovery from stress). The three HRV domains will be assessed at baseline, mid-treatment, and immediately following treatment. Tonic HRV is assessed each week before and after the mindfulness group.
Addiction Cycle Domains in Daily Life | Measured 3x daily
  The negative emotionality domain of the addiction cycle is characterized by temptation to drink in situations when the person is experiencing negative emotions. The Negative Emotionality Scale consists of 2 items scored on a scale from 1=not at all tempted to 5=extremely tempted to drink when experiencing negative emotions. The incentive salience domain of the addiction cycle is characterized by temptation to drink in situations when the person is experiencing rewarding or social pressure to drink. The Incentive Salience Scale consists of 2 items scored on a scale from 1=not at all tempted to 5=extremely tempted to drink when experiencing rewarding, craving, or social situations. The executive function domain of the addiction cycle is characterized by loss of control over drinking. The Executive Scale consists 2 items scored on a scale from 1=indicating more control over drinking to 5=indicating loss. These ecological momentary assessment adapted scales will be delivered 3x per day.

SECONDARY OUTCOMES:
PROMIS Alcohol Negative Consequences | Change between baseline and 6-month follow-up
  The Patient-Reported Outcomes Measurement Information System (PROMIS®) includes 7 items scored from never=1 to almost always=5 that assess negative consequences from alcohol use (e.g., I used poor judgment when I drank). The PROMIS Negative Alcohol Consequences measure will be administered once at baseline, and at follow-up months 3 and 6. Higher scores indicate more negative consequences.
Penn Alcohol Craving Scale | Change from baseline to 6-month follow-up/ 3x daily
  Five item measure of overall craving for alcohol. Responses range from 0 to 6 where 0 represents the absence of the specific craving symptom in the item, and 6 represents the maximum intensity or frequency of the craving symptom in the item. The Penn Alcohol Craving Scale will be administered once at baseline, and at follow-up months 3 and 6. Higher scores on the Penn Alcohol Craving Scale reflect more severe alcohol craving.
  An adapted version of the craving scale will be used 3x daily to assess momentary craving
Reduction in percent heavy drinking days | Change from baseline to 6-month follow-up
  Percent heavy drinking days will be calculated using the Timeline Follow-Back calendar method of assessing standard alcohol drinks consumed each day over the past 90 days. This measure will be used to identify the total number of occasions of daily heavy drinking (defined as 4 or more drinks for females and 5 or more drinks for males), and the percent heavy drinking days will be calculated as the number of heavy drinking days in the past 90 days divided by the total number of days in that time period (typically 90 days, unless some days are missing). The Timeline Follow-Back Calendar will be administered once at baseline, and at follow-up months 3 and 6. Higher percent heavy drinking days indicate more heavy drinking occasions in a 90-day period.
Reduction in drinks per drinking day | Change from baseline to 6-month follow-up
  Drinks per drinking day will be calculated using the Timeline Follow-Back calendar method of assessing standard alcohol drinks consumed each day over the past 90 days. This measure will be used to identify the total number of drinks consumed on each drinking day, and the number of drinks per drinking drinking days will be calculated as the total number of drinks consumed in the past 90 days divided by the total number of days in that time period when drinking occurred (typically 90 days, unless some days are missing). The Timeline Follow-Back Calendar will be administered once at baseline, and at follow-up months 3 and 6. Higher drinks per drinking day indicates greater intensity of drinking in a 90-day period.
Daily drinking quantity and frequency | 3x daily during 8-week intervention period
  The frequency and quantity of drinking will be assessed 3x daily during the 8-week intervention period. A binary outcome of a drinking episode will be used to assessed drinking frequency each day. Quantities will be assessed by asking how many standard drinks the person had (if they reported drinking between assessment periods).

CONTACTS AND LOCATIONS:
Overall Officials: Matison W McCool, Phd, Principal Investigator — Center on Alcohol, Substance use, And Addictions - The University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will comply with all NIAAA Data Archives policies established during the project period. This includes compliance with the NIAAA central data platform requirements and timelines developed through the NIAAA Data Share.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: At the time of publication of the primary manuscript, or within 12 months of last patient assessment.
Access Criteria: mplementation of the plan will follow the NIAAA Data Archive and Data Sharing Policy
URL: https://www.niaaa.nih.gov/research/data-archive-and-resources/niaaa-data-archive